CLINICAL TRIAL: NCT05572255
Title: A Randomized, Open-label, Three-way Crossover Study to Evaluate the Relative Bioavailability of 200 Mg Cenobamate Administered Orally As a Crushed Tablet or a Crushed Tablet Via a Naso-gastric Tube Compared with an Intact 200 Mg Cenobamate Tablet
Brief Title: A Randomized, Open-label, Three-way Crossover Study to Evaluate the Relative Bioavailability of 200 Mg Cenobamate Administered Orally
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YKP3089C045
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Cenobamate

STUDY DESIGN:
Intervention Model Description: Single-dose, 6-sequence, 3-period, 3-treatment crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment A (Reference) (Experimental): An intact 200 mg cenobamate tablet administered orally.
  Interventions: Drug: Cenobamate
- Treatment B (Test 1) (Experimental): A crushed 200 mg cenobamate tablet in suspension administrated orally.
  Interventions: Drug: Cenobamate
- Treatment C (Test 2) (Experimental): A crushed 200 mg cenobamate tablet in suspension administered via an NG tube
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — 200 mg Cenobamate Tablet
  Other Names: YKP3089C045

SUMMARY:
This study is a phase 1, randomized, open-label, single center, single-dose, 6-sequence, 3-period, 3-treatment crossover study in healthy adult male and female subjects to assess: the relative bioavailability of a crushed 200 mg, intact (whole) 200 mg and crushed 200 mg tablet via NG tube of cenobamate. All treatments will be administered under fasting conditions.

DETAILED DESCRIPTION:
This study is a phase 1, randomized, open-label, single center, single-dose, 6-sequence, 3- period, 3-treatment crossover study in healthy adult male and female subjects to assess: the relative bioavailability of a crushed 200 mg cenobamate table in suspension administrated orally (Treatment B, Test 1) compared to an intact (whole) 200 mg cenobamate tablet administered orally (Treatment A, Reference), and the relative bioavailability of a crushed 200 mg cenobamate tablet in suspension administered via an NG tube (Treatment C, Test 2) versus an intact (whole) 200 mg cenobamate tablet (Treatment A, Reference). All treatments will be administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of 18 to 50 years of age (inclusive), at the time of screening
2. Able to read, understand, sign, and date a written informed consent form (ICF) before study participation at screening
3. Agree to use effective methods of contraception as described
4. Body mass index (BMI) between 18.5 and 30.0 kg/m2 (inclusive) at screening
5. In good health on the basis of medical history, physical examination, and routine laboratory measurements (i.e., without clinically relevant pathology)
6. Electrocardiogram (ECG) (12-lead), arterial blood pressure, and heart rate within the normal range of the study center or considered not clinically significant by the Investigator.
7. Able to understand and comply with protocol requirements and instructions and likely to complete the study as planned
8. Females of non-childbearing potential who have undergone a surgical sterilization procedure at least 6 months prior to dosing with official documentation (e.g., bilateral tubal ligation or bilateral salpingectomy or hysterectomy), or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per Principal Investigator's judgment

Exclusion Criteria:

1. Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at Screening that the Investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer.
2. History of nasal obstructions or nasal allergies
3. Smokers, including vaping (subjects who have smoked within 6 months at screening)
4. History of any drug related hypersensitivity reactions as well as severe hypersensitivity reactions (like angioedema) or DRESS as evaluated by the Investigator
5. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with pharmacokinetics of the study drug (except appendectomy and simple hernia repair)
6. Any prescribed or over-the-counter medication taken within 2 weeks prior to start of administration of study drug (Day 1) or within 6 times the elimination half-life of the prescribed or over-the-counter medication prior to start of study drug intake (whichever is longer). Occasional use of acetaminophen is allowed up until 24 hours before dosing
7. Consumption of herbal medications, dietary supplements, and specific fruit products. Subjects should have stopped consumption of herbal medications or dietary supplements (e.g., St. John's Wort, ginkgo biloba, and garlic supplements), and grapefruit or grapefruit juice, or Seville oranges at least 2 weeks before the first dosing day of study drug. Vitamins/mineral supplements are allowed up until 24 hours before dosing
8. History of drug or alcohol abuse or addiction within 2 years before the start of study drug dosing, or a positive test results for alcohol or drugs of abuse, such as amphetamine, barbiturate, benzodiazepine, cocaine, methadone, opiates, oxycodone, phencyclidine, propoxyphene, cannabinoid (THC), MDMA (Ecstasy), cotinine, and tricyclic antidepressant (TCA)
9. Regular consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 pint [473 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) before screening
10. Consumption of an average of more than 5 servings (8 ounces per serving) per day of coffee, cola, or other caffeinated or methyl xanthine beverages before screening
11. Consumption of any caffeine- or methyl xanthine-containing products (e.g., coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours prior to Day 1 of each period and until the end of each PK sampling period
12. Participation in a clinical study involving administration of either an investigational or a marketed drug within 2 months or 7 half-lives (whichever is longer) before screening
13. Blood donation or a significant loss of blood within 60 days of the start of study drug dosing or donation of more than 1 unit of plasma within 7 days before screening
14. Positive result at screening for any of the following infectious disease tests: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antigen and antibody (HIV Ag, HIV Ab)
15. Illness within 5 days before the start of study drug dosing ("illness" is defined as an acute [serious or non-serious] condition [e.g., the flu or the common cold])
16. History of any known relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
17. History of Familial Short QT syndrome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 38 days
  Maximum observed plasma concentration
AUClast | up to 38 days
  AUC from the time 0 to the time of last measurable concentration
AUCinf (AUC0-inf) | up to 38 days
  AUC from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Safety and Tolerability - Adverse Events | up to 45 days
  Number of participants with adverse events (AEs)
Safety and Tolerability - Clinical Laboratory Tests | up to 45 days
  Number of participants with clinical laboratory tests including clinical chemistry, hematology, coagulation, and urinalysis.
Safety and Tolerability - Vitals Signs | up to 45 days
  Number of participants with vitals signs including systolic and diastolic blood pressure, pulse rate, respiratory rate, and body temperature
Safety and Tolerability - Physical Examination | up to 45 days
  Number of participants with physical examination
Safety and Tolerability - ECG | up to 45 days
  Number of participants with ECG QT and RR Intervals
Safety and Tolerability - Columbia Suicide Severity Rating Scale | up to 45 days
  Number of participants with Columbia Suicide Severity Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Vijaykumar Vashi, Study Director — SKLSI
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No